CLINICAL TRIAL: NCT06026462
Title: A Retrospective Cohort Study on the Risk Factors and Prognosis of Asthma With Frequent Acute Attacks Phenotype
Brief Title: Retrospective Cohort Study on Asthma With Frequent Acute Attacks Phenotype
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Liang Dong, Clinical Professor, Qianfoshan Hospital
Other Study IDs: 2022-09-21-03
Record Dates: First submitted 2023-03-28; First posted 2023-09-07 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma with frequent acute exacerbations phenotype: Asthma with frequent acute exacerbations phenotype was defined as having at least two acute attacks in the past 12 months.
  Interventions: Diagnostic Test: Observation of clinical indicators related to asthma
- Asthma with Intermittent acute exacerbations phenotype: Asthma with Intermittent acute exacerbations phenotype was defined as having less than or equal to one acute attacks in the past 12 months.
  Interventions: Diagnostic Test: Observation of clinical indicators related to asthma

INTERVENTIONS:
Diagnostic Test: Observation of clinical indicators related to asthma — Observe the severity of asthma, drug compliance, comorbidities, asthma control, pulmonary function, FeNO, and the number of acute episodes of asthma

SUMMARY:
1. Identify the risk factors for frequent acute exacerbations of asthma: establish a retrospective study, classify patients into frequent acute exacerbation group and non-frequent acute exacerbation group based on the number of acute exacerbations, analyze the characteristics of the two groups, provide clinical, pathological, and comorbidity features of the frequent acute exacerbation subtype of asthma, determine the risk factors associated with frequent acute exacerbations, and establish a disease prediction model for frequent acute exacerbations of asthma.
2. Observe the prognosis and treatment outcome of patients with frequent acute exacerbations of asthma, clarify the relevant factors for poor prognosis in this group of patients, and explore individualized treatment plans to improve the prognosis of patients.
3. Investigate the inflammatory mechanism of frequent acute exacerbations of asthma: use omics methods to screen for subtype-specific biomarkers of frequent acute exacerbations and validate them, clarify the pathogenesis of this subtype, and discover new specific treatment targets.

ELIGIBILITY:
Inclusion Criteria:

18-65 years old, taking asthma medication for at least 4 weeks. The diagnostic criteria for asthma are based on the recommendations of the current guidelines (Guidelines for the Prevention and Treatment of Bronchial Asthma (Version 2020), as follows:

1. Repeated episodes of wheezing, shortness of breath, chest tightness, or coughing are often associated with exposure to allergens, cold air, physical and chemical stimuli, viral upper respiratory tract infections, and exercise.
2. During the attack, scattered or diffuse wheezing sounds can be heard in both lungs, mainly in the expiratory phase, and the expiratory phase is prolonged.
3. The above symptoms and signs can be alleviated by treatment or spontaneously.
4. Except for wheezing, shortness of breath, chest tightness, and coughing caused by other diseases.
5. Those with atypical clinical manifestations (such as no obvious wheezing or physical signs) should have at least one positive pulmonary function test as follows: 1. Positive bronchial provocation test or exercise provocation test; The positive FEV1 of bronchodilator test increased by ≥ 12%;, And the absolute value of FEV1 increase ≥ 200ml; 3. Peak expiratory flow (PEF) intraday (or 2-week) variability ≥ 20%.

Asthma can be diagnosed if it meets the criteria of 1-4 or 4-5.

Exclusion Criteria:

1. Complicated with pneumonia, pulmonary interstitial fibrosis, active pulmonary tuberculosis, obstructive sleep apnea hypopnea syndrome, and other respiratory system related diseases, with a previous history of lung surgery;
2. Those with the following diseases or conditions: severe, progressive, or uncontrolled cardiovascular, liver, kidney, hematopoietic, and neurological disorders; Malignant tumor; Or the presence of immunosuppression (including the use of immunosuppressants or HIV infection resulting in low immune function);
3. Accompanied by severe gastrointestinal diseases (such as inflammatory bowel disease [IBD] or irritable bowel syndrome [IBS]), severe diarrhea (watery stools more than 3 times and lasting for more than 3 days) and constipation (less than 2 stools per week and accompanied by difficulty in defecation) in the past 3 weeks;
4. Systematic application of antibiotics, systemic glucocorticoids (including oral, intravenous [IV] or intramuscular [IM]), microecological agents, or traditional Chinese medicine within the past 4 weeks;
5. Excessive obesity (BMI>32.0 kg/m2), pregnant and lactating women;
6. Poor compliance, unable to cooperate with clinical observation and specimen collection.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Asthma patients who continuously visit our hospital
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Annualized asthma exacerbation rate | one year
  Annual asthma exacerbation rate is calculated as total number of exacerbations of interest divided by the total time at risk

SECONDARY OUTCOMES:
Post-bronchodilator forced expiratory volume in 1 second | up to one year
  Lung function will be described.
Median inhaled corticosteroids (ICS) dose change | one year
  Asthma related ICS use will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Dong, PHD, Principal Investigator — Department of Respiratory and Critical Care Medicine, Shandong Provincial Qianfoshan Hospital